CLINICAL TRIAL: NCT01554540
Title: Pharmacodynamic and Pharmacokinetic Assessment of Treprostinil Iontophoresis on the Forearm and the Fingers
Brief Title: Treprostinil Iontophoresis : a Pharmacodynamic and Pharmacokinetic Study
Acronym: TIPPS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCIC TIPPS 11 18
Record Dates: First submitted 2012-02-07; First posted 2012-03-15 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Scleroderma, Systemic
Keywords: Treprostinil; Scleroderma; Iontophoresis
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cutaneous iontophoresis of Treprostenil (Experimental)
  Interventions: Drug: Cutaneous iontophoresis of treprostinil
- Cutaneous iontophoresis of placebo (Placebo Comparator)
  Interventions: Drug: Cutaneous iontophoresis of treprostinil

INTERVENTIONS:
Drug: Cutaneous iontophoresis of treprostinil — Cutaneous iontophoresis of treprostinil 0.1mg/ml, on the forearm and the fingers. (charge 40-240 mC).

SUMMARY:
The purpose of the study is to assess skin blood flow after non-invasive local administration of treprostinil by using a low-intensity current (i.e. iontophoresis) on the forearm and the fingers of healthy volunteers and patients with systemic sclerosis. The investigators also aim at assessing the systemic bioavailability and dermal diffusion of treprostinil iontophoresis.

DETAILED DESCRIPTION:
Digital ulcerations are a complication of systemic sclerosis (SSc). Available treatments (i.e. IV iloprost) induce major adverse effects, limiting the use of such therapies. Iontophoresis is a non invasive route of administration of drugs. In experimental and clinical preliminary studies, the investigators have shown that iontophoresis of treprostinil on the forearm of healthy subjects induces a sustained increase in skin blood flux and that it is well tolerated (clinicaltrials.gov NCT01082484, manuscript in press). The investigators therefore aim at validating this proof of concept on the digits of SSc patients.

ELIGIBILITY:
Inclusion Criteria:

* Cutaneous systemic scleroderma with sclerosed fingers

Exclusion Criteria:

* pregnant or breast-feeding women
* any chronic disease (in the control group)
* smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-10 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of cutaneous blood flow | 0, 15min, 30 min, 1h, 2h, 4h, 6h, 8h, 10h
  Cutaneous blood flow assessed with Laser Speckle Contrast Imaging (LSCI)

SECONDARY OUTCOMES:
Treprostinil blood concentration | 0, 15min, 30 min, 1h, 2h, 4h, 6h, 8h, 10h
  AUC of treprostinil concentration from the end of iontophoresis until 10 hours after iontophoresis
Treprostinil dermal concentration | 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h
  AUC of treprostinil concentration in the dermis (collected with microdialysis) from the end of iontophoresis until 10 hours after iontophoresis

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Cracowski, MD, Principal Investigator — INSERM 003
Locations (1):
- CIC pharmacology - University Hopsital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Blaise S, Roustit M, Millet C, Ribuot C, Boutonnat J, Cracowski JL. Cathodal iontophoresis of treprostinil and iloprost induces a sustained increase in cutaneous flux in rats. Br J Pharmacol. 2011 Feb;162(3):557-65. doi: 10.1111/j.1476-5381.2010.01045.x. PMID 20860718
- [Background] Cracowski JL, Minson CT, Salvat-Melis M, Halliwill JR. Methodological issues in the assessment of skin microvascular endothelial function in humans. Trends Pharmacol Sci. 2006 Sep;27(9):503-8. doi: 10.1016/j.tips.2006.07.008. Epub 2006 Jul 31. PMID 16876881
- [Background] Herrick AL. Vascular function in systemic sclerosis. Curr Opin Rheumatol. 2000 Nov;12(6):527-33. doi: 10.1097/00002281-200011000-00009. PMID 11092203
- [Background] Kalia YN, Naik A, Garrison J, Guy RH. Iontophoretic drug delivery. Adv Drug Deliv Rev. 2004 Mar 27;56(5):619-58. doi: 10.1016/j.addr.2003.10.026. PMID 15019750
- [Background] Murray AK, Moore TL, King TA, Herrick AL. Vasodilator iontophoresis a possible new therapy for digital ischaemia in systemic sclerosis? Rheumatology (Oxford). 2008 Jan;47(1):76-9. doi: 10.1093/rheumatology/kem314. PMID 18077494
- [Derived] Gaillard-Bigot F, Roustit M, Jourdil JF, Stanke-Labesque F, Cracowski JL. Vascular Effects of Treprostinil Cutaneous Iontophoresis on the Leg, Finger, and Foot. J Clin Pharmacol. 2017 Sep;57(9):1215-1220. doi: 10.1002/jcph.898. Epub 2017 Apr 7. No abstract available. PMID 28387950